CLINICAL TRIAL: NCT00189813
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Potential Efficacy, Safety and Tolerability of Different Oral Doses of YM060 in Patients With Diarrhea-predominant Irritable Bowel Syndrome
Brief Title: A Study of YM060 in Diarrhea-predominant Irritable Bowel Syndrome (d-IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 060-CL-305
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Diarrhea; Nasea®; Irribow®; ramosetron
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea | interventions — ramosetron

INTERVENTIONS:
Drug: YM060

SUMMARY:
This study will examine the efficacy, safety and tolerability of different oral dose of YM060, 5-HT3 receptor antagonist, in patients with d-IBS.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets Rome II criteria for IBS and the subgroup of diarrhea predominant IBS

Exclusion Criteria:

* Patient with severe cardiovascular disease, respiratory diseases, renal diseases, hepatic diseases, digestive tract diseases (excluding IBS), blood diseases, or neurological or psychiatric diseases
* Patient reported having any Type 1 or Type 2 stool on the Bristol Stool Form Scale during the run-in period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 691 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Verbeeck, Study Chair — Director of Late Phase Development
Locations (45):
- Bulgaria (3):
  - Plovdiv
  - Sofia
  - Varna
- Czechia (6):
  - České Budějovice
  - Hradec Králové
  - Ostrava Hrabuvka
  - Prague
  - Tábor
  - Ústí nad Orlicí
- Estonia (3):
  - Tallinn
  - Tartu
  - Viljandi
- Germany (14):
  - Berlin
  - Bochum
  - Dietzenbach
  - Essen
  - Frankfurt
  - Friedberg
  - Hamburg
  - Haßloch
  - Königstein
  - Leipzig
  - Mainz
  - Marburg
  - Potsdam
  - Waltershausen
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Krakow
  - Leszno
  - Lublin
  - Oława
  - Warsaw
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Yaroslavl
- Ukraine (6):
  - Dnipropetrovsk
  - Kiev
  - Lviv
  - Odesa
  - Simferopol
  - Sumy